CLINICAL TRIAL: NCT04593563
Title: The Safety and Efficacy of Psilocybin in Cancer Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maryland Oncology Hematology, PA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49347
Record Dates: First submitted 2020-09-09; First posted 2020-10-20 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder
Keywords: Cancer; Major Depressive Disorder; psychedelics; Psilocybin
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin 25mg (Experimental): Psilocybin 25mg Single does with supportive conditions.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Single 5 capsule oral psilocybin dose: 25mg: 5 x 5 mg capsules.

SUMMARY:
This is a Phase II, single-center, fixed dose, open label trial to explore the safety, tolerability and efficacy of a 25mg dose of psilocybin in cancer patients with MDD. The study population will include adult men and women, 18 years of age or above, with MDD, diagnosed with a malignant neoplasm. MDD is defined as those who meet DSM 5 diagnostic criteria for a single or recurrent episode of MDD without psychotic features. A diagnosis of a malignant neoplasm is defined as having a diagnostic code from C00 to C97 according to the ICD-10.

DETAILED DESCRIPTION:
Recent randomized, placebo-controlled clinical trials of psilocybin therapy for anxiety and depression associated with cancer diagnosis showed significant improvement in study endpoints reflecting psychological distress, as compared to placebo. The effects of a single psilocybin therapy session endured for up to six months with no specific follow-up care. In this study, we aim to explore the safety and efficacy of psilocybin therapy in cancer patients, diagnosed with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. 18 years of age or above at Screening (V1)
3. Currently meet criteria for MDD (single or recurrent episode as defined by DSM 5; if single episode, duration of more or equal to 3 months) based on medical records, clinical assessment and documented completion of the MINI version 7.0.2
4. A diagnosis of a malignant neoplasm with a diagnostic code from C00 to C97 according to the International Classification of Diseases and Related Health Problems, 10th Revision (ICD-10)
5. HAM D 17 score ≥18 at Screening (V1) and at Baseline (V2)
6. Are not currently taking any antidepressant and/or antipsychotic medications, or medical cannabis, at Screening (V1)
7. Able to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits
8. Has capacity to consent (assessed via investigator judgement)

Exclusion Criteria:

Psychiatric Exclusion Criteria:

1. Current or past history of schizophrenia, psychotic disorder, bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history and a structured clinical interview (MINI version 7.0.2)
2. Current (within the past year) alcohol or drug use disorder as defined by DSM 5 (MINI 7.0.2) at Screening (V1)
3. Significant suicide risk as defined by (1) suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year, at Screening or at Baseline, or; (2) suicidal behaviors within the past year, or; (3) clinical assessment of significant suicidal risk during subject interview
4. Other personal circumstances and behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin

   General Medical Exclusion Criteria:
5. Women who are pregnant, nursing, or planning a pregnancy. Women and men of child bearing potential and who are sexually active must agree to use an acceptable contraceptive method throughout their participation in the study. Women of child bearing potential must have a negative urine pregnancy test at Screening (V1) and Baseline (V2)
6. Cardiovascular conditions: recent stroke (<1 year from signing of ICF), recent myocardial infarction (<1 year from signing of ICF), uncontrolled hypertension (blood pressure >140/90) or clinically significant arrhythmia within 1 year of signing the ICF
7. Uncontrolled or insulin dependent diabetes
8. Seizure disorder
9. Positive urine drug screen for illicit drugs or drugs of abuse at V1 and V2. Any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion in conjunction with the medical monitor
10. Current enrollment in any investigational drug or device study or participation in such within 30 days of Screening.
11. Abnormal and clinically significant results on the physical examination, vital signs, ECG, or laboratory tests at Screening (V1) that in the investigator's opinion may consistute a risk for an individual who is explosed to psilocybin. This includes platelets below 50,000 platelets per cubic millimeter of blood, liver function tests three times the upper limit of normal, creatine two times above the normal range. Clinically significant abnormal electrolytes or low hemoglobin (below 8 g/L) should be corrected and rechecked
12. Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study
13. Use of psychedelics, including psilocybin but excluding medical marijuana, within the past 12 months and use of psychedelics during the current episode of depression
14. Concurrent or recent chemotherapy or radiation therapy, that impairs general level of phsyical functioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The Montgomery-Åsberg Depression Rating Scale (MADRS) | 8 weeks
  Ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
  Minimum Score: 0 Maximum Score: 60 Higher Score is indicative of greater depression
Quick Inventory of Depressive Symptomatology Self reported (QIDS-SR) | 8 weeks
  16-Item quick inventory of depressive symptomatology. Minimum score: 0 Maximum Score: 16 Higher Score is indicative of worsening depression.
Maudsley Visual Analogue Scale (VAS) current | 8 weeks
  Minimum score: -50 Maximum Score: 50 Higher score is indicative of a better outcome.
Maudley Visual Analogue Scale (VAS) Change. | 8 weeks
  Change in Maudsley VAS change scores from Baseline Minimum score: -50 Maximum Score: 50 Higher score is indicative of a better outcome.
Pain Visual Analogue Score (VAS) | 8 weeks
  Change in use of pain medications from Baseline (Day -1 [V2]) to Week 8 (V7) Minimum score: 0 Maximum Score: 10 Higher score is not indicative of a better outcome.
Hamilton Anxiety Rating Scale-A (HAM-A) | 8 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) is a widely used and well-validated tool for measuring the severity of a patient's anxiety. It should be administered by an experi- enced clinician. The HAM-A probes 14 parameters and takes 15-20 minutes to complete the interview and score the results. Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe.
  Minimum Score: 0 Maximum Score: 56 Higher Score is indicative of worsening Depression
State-Trait Anxiety Inventory (STAI) | 8 weeks
  Psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis Minimum: 20 Maximum: 80 Higher Score is indicative of worsening outcome.
National Institute of Health Healing Experience of All Life Stressors (NIH-HEALS) | 8 weeks
  Psycho-social-spiritual healing in NIH-HEALS total score change from Baseline (Day -1 [V2]) to Weeks 1 (V5), 3 (V6), and 8 (V7). Additionally changes in the three factor scores on this measure will be assessed for change at the same timepoints: Connection; Reflection and Introspection; Trust and Acceptance.Healing Experience of All Life Stressors (NIH-HEALS) was developed by the NIH Clinical Center Pain and Palliative Care Service as a psycho-social-spiritual measure of healing that assesses positive transformation in response to challenging life events. It is a self-report, 35-item questionnaire.
Patient EQ-5D-5L | 8 weeks
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Participant EQ 5D 5L score change from Baseline (Day -1 [V2]) to subsequent follow up visits.
  Minimum: 0 Maximum: 20 Higher Score is indicative of worsening outcome.
Caregiver Oncology Quality of Life Questionnaire (CarGOQol) | 8 weeks
  CarGOQol score change from Baseline (Day -1 [V2]) to subsequent follow up visits (this assessment is not mandatory) Minimum: 0 Maximum: 116 Higher Score is indicative of worsening outcome.
DS-II | 8 weeks
  Change in DS-II factor scores from Baseline. Minimum: 0 Maximum: 32 Higher Score is indicative of worsening outcome.
5 Dimension Altered State of Consciousness (5D-ASC) | 8 weeks
  Summary of the 5D-ASC on the day of psilocybin dosing. o Links between psychedelic intensity and experience (via the 5D-ASC) and depression and anxiety outcomes will also be explored and patient experience and acceptability of the treatment summarised at V3 and V4.
  This has 11 subscales, and higher scores are indicative of good outcomes.
Sheehan Disability Score (SDS) | 8 weeks
  SDS score change from Baseline Minimum: 0 Maximum: 30 Higher Score is indicative of worsening outcome.
Scale To Assess Therapeutic Relationship: Patient (STAR-P) | 8 weeks
  Therapeutic alliance of the clinician and patient, as rated using the STAR-C and STAR-P respectively will be assessed at Baseline, along with assessing correlations with this measure and primary and secondary outcomes as a possible predictor of response Minimum: 0 Maximum: 48 Higher Score is indicative of good outcome.
Scale To Assess Therapeutic Relationship: Clinician. (STAR-C) | 8 weeks
  Therapeutic alliance of the clinician and patient, as rated using the STAR-C and STAR-P respectively will be assessed at Baseline, along with assessing correlations with this measure and primary and secondary outcomes as a possible predictor of response Minimum: 0 Maximum: 48 Higher Score is indicative of good outcome.
Changes in electrocardiographs. | 8 weeks
  Abnormal and clinically significant results on the ECG, that in the investigator's opinion may constitute a risk for an individual who is exposed to psilocybin.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Oncology Hematology PA, Rockville, Maryland, United States

REFERENCES:
- [Derived] Agrawal M, Richards W, Beaussant Y, Shnayder S, Ameli R, Roddy K, Stevens N, Richards B, Schor N, Honstein H, Jenkins B, Bates M, Thambi P. Psilocybin-assisted group therapy in patients with cancer diagnosed with a major depressive disorder. Cancer. 2024 Apr 1;130(7):1137-1146. doi: 10.1002/cncr.35010. Epub 2023 Dec 18. PMID 38105655